CLINICAL TRIAL: NCT00300612
Title: A Phase I/II Study of Dorgenmeltucel-L (HyperAcute Melanoma) an Antitumor Vaccination Using Alpha(1,3)Galactosyltransferase Expressing Allogeneic Tumor Cells in Patients With Refractory or Recurrent Malignant Melanoma
Brief Title: Vaccine Treatment for Advanced Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Nicholas N. Vahanian, M.D., Chief Medical and Operations Officer, NewLink Genetics Corporation
Organization: Lumos Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0104; OBA#0404-640
Record Dates: First submitted 2006-03-07; First posted 2006-03-09 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vaccine group (Experimental)
  Interventions: Biological: HyperAcute-Melanoma Vaccine

INTERVENTIONS:
Biological: HyperAcute-Melanoma Vaccine — Cells will be injected intradermally every two weeks for twelve vaccinations. If the patient completes all twelve vaccinations, dosage will vary from a total of 1.3 x 109 to 3.8 x 109 HyperAcute™-Melanoma Vaccine cells administered.
  Other Names: HAM-1, HAM-2, and HAM-3

SUMMARY:
This 2-phase study will determine the safety of treating patients with malignant melanoma with the genetically engineered HyperAcute-Melanoma vaccine. It will establish the proper vaccine dose and will examine side effects and potential benefits of the treatment. The vaccine contains killed melanoma cells containing a mouse gene that causes the production of a foreign pattern of protein-sugars on the cell surface. It is hoped that the immune response to the foreign substance will stimulate the immune system to attack the patient's own cancer cells that have similar proteins without this sugar pattern, causing the tumor to remain stable or shrink.

Patients 18 years of age or older with malignant melanoma may be eligible for this study. Candidates will be screened with medical history and physical examination, blood tests, urinalysis, chest x-rays and CT scans. MRI, PET, and ultrasound scans may be obtained if needed.

Participants will receive twelve vaccinations two weeks apart from each other. The vaccines will be injected under the skin, similar to the way a tuberculosis skin test is given. Phase I of the study will treat successive groups of patients with increasing numbers of the vaccine cells to evaluate side effects of the treatment and determine the optimum dose. Phase II will look for any beneficial effects of the vaccine given at the highest dose found to be safe in Phase I. Monthly blood samples will be drawn during the 6 months of vaccine treatment. In addition, patient follow-up visits will be scheduled every 3 months for the remaining first year (6 months) after vaccination and then every 6 months for the next 2 years for the following tests and procedures to evaluate treatment response and side effects:

Medical history and physical examination Blood tests X-rays and various scans (nuclear medicine/CT/MRI) FACT-G Assessment questionnaire to measure the impact of treatment on the patient's general well-being. The questionnaire is administered before beginning treatment, monthly during treatment, and during follow-up visits after completing the treatment. It includes questions on the severity of cancer symptoms and the ability to perform normal activities of daily life.

DETAILED DESCRIPTION:
According to statistics of the American Cancer Society, an estimated 55,000 individuals will be diagnosed with malignant melanoma and 8,000 will die of the disease this year in the Unites States despite all current therapy. This protocol attempts to exploit an approach to melanoma vaccine therapy using a naturally occurring barrier to xenotransplantation in humans in attempt to vaccinate patients against their melanoma The expression of the murine alpha(1,3)galactosyltransferase [alpha(1,3)GT] gene results in the cell surface expression of alpha(1,3)galactosyl-epitopes (alpha-gal) on membrane glycoproteins and glycolipids. These epitopes are the major target of the hyperacute rejection response that occurs when organs are transplanted from non-primate donor species into man. Human hosts often have pre-existing anti-alpha-gal antibodies that bind alpha-gal epitopes and lead to rapid activation of complement and cell lysis. The pre-existing anti-alpha-gal antibodies found in most individuals are thought to be due to exposure to alpha-gal epitopes that are naturally expressed on normal gut flora leading to chronic immunological stimulation. These antibodies may comprise up to 1% of serum IgG. In this Phase I/II trial, patients with advanced stage melanoma will undergo a series of twelve intradermal injections with a trivalent vaccine composed of irradiated allogeneic melanoma cell lines (HAM-1, HAM-2 and HAM-3). These cell lines have been transduced with a recombinant Moloney murine leukemia virus (MoMLV)-based retroviral vector expressing the murine alpha(1,3)GT gene. Endpoints of the study include determination of dose-limiting toxicity (DLT), maximum tolerated dose (MTD), tumor and immunological responses.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of malignant melanoma. (pathology must be reviewed by Pathology Department)
* AJCC Stage IIIC (any T, N1b, N2b, N3, M0) or Stage IV (any T, any N, M1), metastatic, progressive, refractory, recurrent, or high risk of recurrence malignant melanoma.
* Adult patients > or = to 18 years of age
* Measurable or non-measurable disease.
* Patient is > or = to 4 weeks past major surgery, radiotherapy, chemotherapy. (6 weeks if treated with a nitrosureas) or biotherapy/targeted therapies and has recovered from the toxicity of prior treatment to < or = to Grade 1, exclusive of alopecia or fatigue.
* Hemoglobin > or = to 10.0 gm/dL, absolute granulocyte count > or = to 1500/ mm3,platelets > or = to 100,000/ mm3, absolute lymphocyte count > or = to 475/ mm3.
* Total Bilirubin < or = to 1.5 ULN (mg/dL), ALT (SGPT) and AST (SGOT) < or = to 2.5 x ULN.
* Serum creatinine < or = to 1.5 x ULN, or creatinine clearance > or = to 50 mL/min.
* Serum albumin > or = to 3.0 gm/dL.
* ECOG performance status < or = to 2.
* All On-Study Test results are < or = to Grade I toxicity for patient to be eligible for study, except for serum LDH. PT, PTT must be < or = to 1.5 x ULN except for patients who are on therapeutic anticoagulant therapy.
* Negative serologies for Hepatitis B, Hepatitis C, and HIV
* Ability to give informed consent and express a willingness to meet all the expected requirements of the protocol including using contraception as outlined in the consent form.
* Expected survival > 6 months. NOTE: Prior therapy for melanoma may include surgery, radiation therapy, immunotherapy including interleukins and interferon, and/or < or = to 2 different chemotherapy regimens and other experimental therapies.

Exclusion Criteria:

* Subject has an active CNS metastases or carcinomatous meningitis. Subjects with CNS lesions that have been treated and show no evidence of progression on CT/MRI for > or = to 3 months are eligible.
* Hypercalcemia > 2.9 mmol/L, unresponsive to standard therapy (IV hydration, diuretics calcitonin and/or bisphosphate therapy)
* Subject is any of the following: HIV positive, history or hepatitis C virus infection, acute or chronic active hepatitis B virus infection (HbsAg positive).
* Subject has had splenectomy.
* Subject has had other malignancy within five years, and probability of recurrence of prior malignancy is >5%. (if less than 5% subject is eligible) SEE NOTE1
* Subject has history of organ transplant or currently taking active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subject is currently receiving systemic corticosteroid therapy for any reason. SEE NOTE2
* Subject has significant or uncontrolled congestive heart failure, myocardial infarction or significant ventricular arrhythmias within the last six months or significant pulmonary dysfunction.
* Subject has an active infection or antibiotics within 1-week prior to study,including unexplained fever (temp > 38.1C)
* Subject has an autoimmune disease (systemic lupus erythematosis, active rheumatoid arthritis, etc.) with the exception of vitiligo. SEE NOTE3.
* Subject has a serious medical condition that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis)
* Subject has any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with an aspect of the study.
* Subject has a known allergy to a component of the alpha(1,3)galactosyltransferase tumor vaccine or cell lines from which it is derived.
* Subject is pregnant or nursing.

NOTE1: Subjects curatively treated for squamous and basal cell carcinoma of the skin and carcinoma in situ of the uterine cervix (CIN) or subjects with a history of malignant tumor in the past that has been disease free for at least five years are also eligible for this study.

NOTE2: Subject's receiving inhaled or topical corticosteroids are eligible. Subjects who require systemic corticosteroid therapy after beginning vaccination will be removed from the study.

NOTE3: Subjects with a remote history of asthma or mild active asthma are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To assess the side effects, dose-limiting toxicity and maximum tolerated dose. | 6 months

SECONDARY OUTCOMES:
To assess tumor response and immunological response. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C. DeConti, M.D., Principal Investigator — University of South Florida; Charles J. Link, M.D., Study Chair — NewLink Genetics Corporation
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States